CLINICAL TRIAL: NCT00003130
Title: Prospective Evaluation of Body Surface Area (BSA) as a Determinant of Paclitaxel Pharmacokinetics/Pharmacodynamics in Women With Solid Tumors
Brief Title: Paclitaxel in Treating Women With Recurrent Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9763; U10CA031946 (NIH); CALGB-9763; CDR0000065893 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-11-25 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paclitaxel (Experimental): Patients receive single fixed dose intravenous paclitaxel over 3 hours on day 1. Blood samples must be drawn prior to the first paclitaxel infusion and then at 1, 6, and 24 hours after the start of the infusion during course 1 only. Treatment courses of intravenous paclitaxel are repeated every 3 weeks at the discretion of the treating physician. Patients are evaluated for response after the second course. Patients are followed at the discretion of the physician.
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating women who have recurrent solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the relationships between body surface area (BSA) and toxic effects, BSA and pharmacokinetics, and pharmacokinetics and toxic effects in women with recurrent solid tumors who receive a fixed total dose of paclitaxel. II. Determine the toxic effects of paclitaxel in these patients. III. Assess the pharmacokinetics of paclitaxel in these patients.

OUTLINE: Patients receive single fixed dose intravenous paclitaxel over 3 hours on day 1. Blood samples must be drawn prior to the first paclitaxel infusion and then at 1, 6, and 24 hours after the start of the infusion during course 1 only. Treatment courses of intravenous paclitaxel are repeated every 3 weeks at the discretion of the treating physician. Patients are evaluated for response after the second course. Patients are followed at the discretion of the physician.

PROJECTED ACCRUAL: A total of 50 patients will be accrued over 13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent adult solid tumors Must have measurable or evaluable disease No known bone marrow metastasis

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Women Performance Status: Zubrod 0-2 Life Expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL SGOT less than 2.0 times upper limit of normal Renal: Creatinine no greater than 1.5 times upper limit of normal Other: Concurrently active secondary malignancies are allowed

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior paclitaxel therapy No more than 1 prior chemotherapy regimen for metastatic disease At least 4 weeks since chemotherapy Greater than 6 weeks since nitrosoureas, melphalan, or mitomycin Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since radiotherapy No prior whole pelvic radiation Surgery: At least 4 weeks since major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 1997-11; Primary Completion 2002-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonius A. Miller, MD, Study Chair — Wake Forest University Health Sciences
Locations (34):
- United States (34):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Miller AA, Rosner GL, Egorin MJ, Hollis D, Lichtman SM, Ratain MJ. Prospective evaluation of body surface area as a determinant of paclitaxel pharmacokinetics and pharmacodynamics in women with solid tumors: Cancer and Leukemia Group B Study 9763. Clin Cancer Res. 2004 Dec 15;10(24):8325-31. doi: 10.1158/1078-0432.CCR-04-1078. PMID 15623609